CLINICAL TRIAL: NCT00233987
Title: Tandem Autologous Stem Cell Transplantation for Patients With Primary Progressive or Recurrent Hodgkin's Disease (A BMT Study), Phase II
Brief Title: S0410 Tandem Stem Cell Transplantation in Treating Patients With Progressive or Recurrent Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000442392; U10CA032102 (NIH); S0410 (Other: SWOG)
Record Dates: First submitted 2005-10-05; First posted 2005-10-06 (Estimated); Results first posted 2013-02-05 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-01

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Carmustine; Cyclophosphamide; Etoposide; Melphalan; Radiotherapy; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- High-dose therapy plus tandem transplant (Experimental): Regimen consists of 2 cycles of high-dose therapy, each followed by stem cell infusion. Cycle 1 consists of high-dose melphalan followed by infusion of approximately 1.5 million cluster of differentiation 34 positive (CD34+) cells. Cycle 2 consists of either TBI-based or 1,3-bis(2-chloroethyl)-1-nitrosourea (BCNU)-based high-dose therapy followed by infusion of at least 2 million CD34+ cells.
  Interventions: Drug: carmustine; Drug: cyclophosphamide; Drug: etoposide; Drug: melphalan; Procedure: autologous-autologous tandem hematopoietic stem cell transplantation; Radiation: radiation therapy

INTERVENTIONS:
Drug: carmustine — 150 mg/m^2 IV over 2 hours 4, 5, and 6 days before transplant.
  Other Names: BCNU
Drug: cyclophosphamide — 100 mg/kg IV 2 days before transplant.
Drug: etoposide — 60 mg/kg IV over 4 hours 4 days before transplant.
Drug: melphalan — 150 mg/m^2 IV 1 day before transplant.
Procedure: autologous-autologous tandem hematopoietic stem cell transplantation — 2.0 x 10^6 CD34+ cells, beginning at least 24 hours after melphalan infusion.
Radiation: radiation therapy — 150 centigray (cGy) total body irradiation given b.i.d on days 5-8 before transplant.
  Other Names: Total body irradiation (TBI)

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill cancer cells. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving chemotherapy with a peripheral stem cell transplant may allow more chemotherapy to be given so that more cancer cells are killed. Tandem (two) autologous stem cell transplants may be an effective treatment for Hodgkin's lymphoma.

PURPOSE: This phase II trial is studying how well tandem stem cell transplantation works in treating patients with progressive or recurrent Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the 2-year progression-free survival of patients with progressive or recurrent Hodgkin's lymphoma treated with tandem autologous stem cell transplantation (2 courses of high-dose therapy with autologous stem cell rescue).
* Determine the response rate in patients treated with this regimen.
* Determine the toxic effects of this regimen in these patients.

OUTLINE: This is a multicenter study.

* Salvage therapy (for patients with relapsed disease after achieving a previous complete response): Patients receive at least 2 courses of salvage chemotherapy or radiotherapy. No more than 6 weeks later, patients proceed to autologous hematopoietic stem cell collection.
* Autologous hematopoietic stem cell collection: Patients undergo autologous hematopoietic stem cell collection. Patients with an inadequate number of collected stem cells are removed from the study.
* Pre-transplant salvage radiation: Patients with residual tumor greater than 5 cm after initial salvage therapy undergo involved-field radiotherapy. All patients then proceed to the first preparative regimen.
* First preparative regimen: Patients receive high-dose melphalan IV on day -1.
* First autologous stem cell transplantation (SCT): Patients undergo autologous SCT on day 0. At least 28 days later, patients proceed to second preparative regimen.
* Second preparative regimen: Patients receive 1 of the following preparative regimens:

  * Total-body irradiation (TBI)-based regimen: Patients undergo TBI twice daily on days -8 to -5. Patients also receive etoposide IV over 4 hours on day -4 and cyclophosphamide IV over 1 hour on day -2.
  * Carmustine-based regimen: Patients receive carmustine IV over 2 hours on days -6 to -4, etoposide IV over 4 hours on day -4, and cyclophosphamide IV over 1 hour on day -2.
* Second autologous SCT: Patients undergo second autologous SCT on day 0. After completion of study treatment, patients are followed every 6 months for 2 years and then annually for up to 7 years.

PROJECTED ACCRUAL: A total of 85 patients will be accrued for this study over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed Hodgkin's lymphoma

  * Relapsed or refractory disease
  * Biopsy or radiological evidence of disease at time of recurrence/progression required
* Has received ≥ 1 prior systemic chemotherapy regimen
* No clonal abnormalities in marrow collection
* Must undergo involved-field radiotherapy if bulky disease > 5 cm
* Must have adequate sections of original diagnostic specimen available for review

  * Needle aspirations or cytologies are not adequate
* No prior lymphoma, myelodysplastic syndromes, or leukemia (even if disease free > 5 years)
* Patients who relapse after achieving a complete remission must complete a minimum of 2 courses of salvage chemotherapy or radiation therapy to determine if sensitive or resistant recurrent disease is present
* No central nervous system (CNS) involvement

PATIENT CHARACTERISTICS:

Age

* 15 to 70

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN) (unless due to Hodgkin's disease)

Renal

* Creatinine clearance ≥ 60 mL/min
* Creatinine ≤ 2 times upper limit of normal

Cardiovascular

* None of the following conditions requiring therapy:

  * Coronary artery disease
  * Cardiomyopathy
  * Congestive heart failure
  * Arrhythmias
* Ejection fraction ≥ 45% by Multi Gated Acquisition Scan (MUGA) or 2-D echocardiogram

Pulmonary

* Adequate pulmonary function
* Corrected diffusing capacity of lung for carbon monoxide (DLCO) ≥ 60% OR
* Forced Expiratory Volume in One Side (FEV_1) ≥ 60% of predicted

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer
* No known HIV or AIDS infection
* No active bacterial, fungal, or viral infection
* No medical condition that would preclude study treatment

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics

Surgery

* Not specified

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2005-10; Primary Completion 2014-11 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eileen P. Smith, MD, Study Chair — City of Hope Comprehensive Cancer Center; Patrick J. Stiff, MD, Study Chair — Loyola University; Louis S. Constine, MD, Study Chair — James P. Wilmot Cancer Center
Locations (53):
- United States (53):
  - University of California Davis Cancer Center, Sacramento, California
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Auburn Regional Center for Cancer Care, Auburn, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington

REFERENCES:
- [Derived] Smith EP, Li H, Friedberg JW, Constine LS, Rimsza LM, Cook JR, Laport GG, Popplewell LL, Holmberg LA, Smith SM, LeBlanc M, Forman SJ, Fisher RI, Stiff PJ. Tandem Autologous Hematopoietic Cell Transplantation for Patients with Primary Progressive or Recurrent Hodgkin Lymphoma: A SWOG and Blood and Marrow Transplant Clinical Trials Network Phase II Trial (SWOG S0410/BMT CTN 0703). Biol Blood Marrow Transplant. 2018 Apr;24(4):700-707. doi: 10.1016/j.bbmt.2017.12.798. Epub 2017 Dec 28. PMID 29289757

RESULTS

PARTICIPANT FLOW:
Groups:
- High-dose Therapy Plus Tandem Transplant: Regimen consists of 2 cycles of high-dose therapy, each followed by stem cell infusion. Cycle 1 consists of high-dose melphalan followed by infusion of approximately 1.5 million CD34+ cells. Cycle 2 consists of either Total Body Irradiation(TBI)-based or 1,3-bis (2-chloroethyl)-1-nitrosourea(BCNU)-based high-dose therapy followed by infusion of at least 2 million cluster of differentiation 34 positive (CD34+) cells.
Period: Overall Study
Arm/Group | High-dose Therapy Plus Tandem Transplant
Started | 98
Eligible | 94
Eligible and Treated | 92
Completed | 83
Not Completed | 15
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 2
Not completed — Reason Under Review | 1
Not completed — Other - Not Protocol Specified | 5
Not completed — Eligible but No Treatment Received | 2
Not completed — Ineligible | 4

BASELINE CHARACTERISTICS:
Groups:
- High-dose Therapy Plus Tandem Transplant: Regimen consists of 2 cycles of high-dose therapy, each followed by stem cell infusion. Cycle 1 consists of high-dose melphalan followed by infusion of approximately 1.5 million CD34+ cells. Cycle 2 consists of either TBI-based or BCNU-based high-dose therapy followed by infusion of at least 2 million CD34+ cells.
Arm/Group | High-dose Therapy Plus Tandem Transplant
Number analyzed (Participants) | 92
Age, Continuous [Median (Full Range); unit: years] | 34.1 [18.2 to 60.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 77
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: 2-year Progression-free Survival
Description: Measured from date of randomization to date of first observation of progressive disease, or death due to any cause
Time Frame: At day 60, then every 6 months for 2 years
Population: All eligible patients who started treatment were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | High-dose Therapy Plus Tandem Transplant
Number analyzed (Participants) | 92
percentage of participants | 59 [49 to 69]

2. Secondary Outcome: Response Rate
Description: Complete Response(CR) is a complete disappearance of all disease with the exception of nodes. No new lesions. previously enlarged organs must have regressed and not be palpable. Bone marrow(BM) must be negative if positive at baseline. Normalization of markers. CR Unconfirmed (CRU) does not qualify for CR above, due to a residual nodal mass or an indeterminate BM. Partial Response(PR) is a 50% decrease in the sum of products of greatest diameters (SPD) for up to 6 identified dominant lesions, including spleenic and hepatic nodules from baseline. No new lesions and no increase in the size of liver, spleen or other nodes.
Time Frame: At day 60, then every 6 months for 2 years
Population: All eligible patients who started treatment were included in the analysis. Five patients with no evidence of disease at baseline were excluded.
Measure: Number; unit: participants
Arm/Group | High-dose Therapy Plus Tandem Transplant
Number analyzed (Participants) | 87
participants
  Complete Response | 15
  Partial Response | 8
  Unconfirmed Complete Response | 3
  Unconfirmed Partial Response | 2
  No Response | 33
  Assessment Inadequate | 26

3. Secondary Outcome: Overall Survival
Description: Measured from date of registration to date of death due to any cause or last contact
Time Frame: At day 60, then every 6 months for 2 years, then annually for a total of 7 years
Population: All eligible patients who started treatment were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | High-dose Therapy Plus Tandem Transplant
Number analyzed (Participants) | 92
percentage of participants | 91 [83 to 95]

4. Secondary Outcome: Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug
Description: Adverse Events (AEs) are reported by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. For each patient, worst grade of each event type is reported. Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Fatal.
Time Frame: Assessed after cycle 1 high dose therapy, after cycle 2 high dose therapy, and at 1 month and 2 months after the second stem cell infusion
Population: Eligible patients who had received any treatment were included in the adverse event summaries. Any CTCAE 3.0 event of Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal) which deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Arm/Group | High-dose Therapy Plus Tandem Transplant
Number analyzed (Participants) | 90
Participants
  ALT, SGPT (serum glutamic pyruvic transaminase) | 6
  AST, SGOT | 4
  Allergic reaction/hypersensitivity | 3
  Anorexia | 20
  Bilirubin (hyperbilirubinemia) | 1
  Calcium, serum-low (hypocalcemia) | 1
  Colitis, infectious (e.g., Clostridium difficile) | 1
  Confusion | 1
  Constitutional Symptoms-Other (Specify) | 1
  Cough | 1
  Dehydration | 6
  Dermatology/Skin-Other (Specify) | 1
  Diarrhea | 8
  Distention/bloating, abdominal | 1
  Dry mouth/salivary gland (xerostomia) | 1
  Dysphagia (difficulty swallowing) | 6
  Dyspnea (shortness of breath) | 5
  Edema: limb | 1
  Esophagitis | 5
  Fatigue (asthenia, lethargy, malaise) | 4
  Febrile neutropenia | 47
  Fever in absence of neutropenia, ANC lt1.0x10e9/L | 3
  Glucose, serum-high (hyperglycemia) | 6
  Hemoglobin | 22
  Hemorrhage, pulmonary/upper respiratory - Nose | 2
  Hemorrhage/Bleeding-Other (Specify) | 1
  Hypotension | 10
  Hypoxia | 4
  Inf (clin/microbio) w/Gr 3-4 neuts - Abdomen NOS | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Blood | 2
  Inf (clin/microbio) w/Gr 3-4 neuts - Catheter-rel | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Foreign body | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Lung | 3
  Inf (clin/microbio) w/Gr 3-4 neuts - Rectum | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Sinus | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Skin | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Stomach | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Upper airway | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Blood | 2
  Inf w/normal ANC or Gr 1-2 neutrophils - Catheter | 1
  Infection with unknown ANC - Blood | 1
  Infection with unknown ANC - Skin (cellulitis) | 1
  Infection-Other (Specify) | 5
  Leukocytes (total WBC) | 65
  Lymphatics-Other (Specify) | 1
  Lymphopenia | 50
  Magnesium, serum-high (hypermagnesemia) | 1
  Mood alteration - depression | 2
  Mucositis/stomatitis (clinical exam) - Oral cavity | 9
  Mucositis/stomatitis (clinical exam) - Pharynx | 8
  Mucositis/stomatitis (functional/symp) - Oral cav | 6
  Mucositis/stomatitis (functional/symp) - Pharynx | 10
  Nausea | 32
  Neutrophils/granulocytes (ANC/AGC) | 67
  Opportunistic inf associated w/gt=Gr 2 lymphopenia | 1
  Pain - Head/headache | 2
  Pain - Joint | 2
  Pain - Oral cavity | 2
  Pain - Throat/pharynx/larynx | 3
  Pain-Other (Specify) | 2
  Phosphate, serum-low (hypophosphatemia) | 25
  Platelets | 70
  Pneumonitis/pulmonary infiltrates | 3
  Potassium, serum-low (hypokalemia) | 13
  Pruritus/itching | 1
  Psychosis (hallucinations/delusions) | 1
  Pulmonary hypertension | 1
  Rash/desquamation | 4
  SVT and nodal arrhythmia - SVT tachycardia | 1
  Sodium, serum-low (hyponatremia) | 11
  Syndromes-Other (Specify) | 2
  Thrombosis/thrombus/embolism | 2
  Uric acid, serum-high (hyperuricemia) | 1
  Vomiting | 12

ADVERSE EVENTS:
Time Frame: Assessed after cycle 1 high dose therapy, after cycle 2 high dose therapy, and at 1 month and 2 months after the second stem cell infusion
Arm/Group | High-dose Therapy Plus Tandem Transplant
Serious Adverse Events (participants affected / at risk) | 2/90
Other Adverse Events (participants affected / at risk) | 88/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High-dose Therapy Plus Tandem Transplant (N=90)
Inf (clin/microbio) w/Gr 3-4 neuts - Catheter-rel (Infections and infestations) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High-dose Therapy Plus Tandem Transplant (N=90)
Febrile neutropenia (Blood and lymphatic system disorders) | 48
Hemoglobin (Blood and lymphatic system disorders) | 68
SVT and nodal arrhythmia - Sinus bradycardia (Cardiac disorders) | 6
SVT and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 33
Ocular/Visual-Other (Specify) (Eye disorders) | 6
Constipation (Gastrointestinal disorders) | 23
Diarrhea (Gastrointestinal disorders) | 66
Distention/bloating, abdominal (Gastrointestinal disorders) | 9
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 17
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 14
Esophagitis (Gastrointestinal disorders) | 13
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 6
Gastrointestinal-Other (Specify) (Gastrointestinal disorders) | 8
Heartburn/dyspepsia (Gastrointestinal disorders) | 31
Hemorrhoids (Gastrointestinal disorders) | 6
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 28
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 14
Nausea (Gastrointestinal disorders) | 82
Pain - Abdomen NOS (Gastrointestinal disorders) | 36
Pain - Oral cavity (Gastrointestinal disorders) | 21
Pain - Rectum (Gastrointestinal disorders) | 10
Pain - Stomach (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 71
Edema: head and neck (General disorders) | 5
Edema: limb (General disorders) | 22
Fatigue (asthenia, lethargy, malaise) (General disorders) | 64
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 36
Pain - Chest/thorax NOS (General disorders) | 11
Pain - Face (General disorders) | 7
Pain-Other (Specify) (General disorders) | 35
Rigors/chills (General disorders) | 38
Allergic reaction/hypersensitivity (Immune system disorders) | 10
Infection-Other (Specify) (Infections and infestations) | 16
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 49
AST, SGOT (Investigations) | 49
Alkaline phosphatase (Investigations) | 26
Bilirubin (hyperbilirubinemia) (Investigations) | 6
Cholesterol, serum-high (hypercholesterolemia) (Investigations) | 7
Creatinine (Investigations) | 18
GGT (gamma-glutamyl transpeptidase) (Investigations) | 5
Leukocytes (total WBC) (Investigations) | 66
Lymphopenia (Investigations) | 53
Metabolic/Laboratory-Other (Specify) (Investigations) | 5
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 69
Platelets (Investigations) | 75
Weight gain (Investigations) | 10
Weight loss (Investigations) | 21
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 56
Anorexia (Metabolism and nutrition disorders) | 53
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 37
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 11
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 54
Dehydration (Metabolism and nutrition disorders) | 7
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 52
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 6
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 6
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 28
Obesity (Metabolism and nutrition disorders) | 5
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 48
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 55
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 43
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 10
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 9
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 18
Pain - Back (Musculoskeletal and connective tissue disorders) | 26
Pain - Bone (Musculoskeletal and connective tissue disorders) | 15
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 10
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 8
Pain - Joint (Musculoskeletal and connective tissue disorders) | 11
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 9
Pain - Neck (Musculoskeletal and connective tissue disorders) | 7
Dizziness (Nervous system disorders) | 32
Neuropathy: sensory (Nervous system disorders) | 13
Ocular/Visual-Other (Specify) (Nervous system disorders) | 6
Pain - Head/headache (Nervous system disorders) | 50
Somnolence/depressed level of consciousness (Nervous system disorders) | 16
Taste alteration (dysgeusia) (Nervous system disorders) | 13
Insomnia (Psychiatric disorders) | 43
Mood alteration - agitation (Psychiatric disorders) | 7
Mood alteration - anxiety (Psychiatric disorders) | 46
Mood alteration - depression (Psychiatric disorders) | 18
Hemorrhage, GU - Urinary NOS (Renal and urinary disorders) | 5
Renal/Genitourinary-Other (Specify) (Renal and urinary disorders) | 8
Urinary frequency/urgency (Renal and urinary disorders) | 5
Hemorrhage, GU - Vagina (Reproductive system and breast disorders) | 5
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 21
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 36
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 20
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 11
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 9
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 9
Mucositis/stomatitis (clinical exam) - Pharynx (Respiratory, thoracic and mediastinal disorders) | 34
Mucositis/stomatitis (functional/symp) - Pharynx (Respiratory, thoracic and mediastinal disorders) | 24
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 31
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 13
Pulmonary/Upper Respiratory-Other (Specify) (Respiratory, thoracic and mediastinal disorders) | 16
Dermatology/Skin-Other (Specify) (Skin and subcutaneous tissue disorders) | 26
Dry skin (Skin and subcutaneous tissue disorders) | 13
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 31
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 11
Pruritus/itching (Skin and subcutaneous tissue disorders) | 17
Rash/desquamation (Skin and subcutaneous tissue disorders) | 35
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 6
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 5
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 14
Flushing (Vascular disorders) | 18
Hemorrhage/Bleeding-Other (Specify) (Vascular disorders) | 7
Hot flashes/flushes (Vascular disorders) | 6
Hypertension (Vascular disorders) | 15
Hypotension (Vascular disorders) | 47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No